CLINICAL TRIAL: NCT06291727
Title: Mepivacaine Versus Bupivacaine Spinal Anesthesia for Same Day Discharge Following Total Knee Arthroplasty
Brief Title: Mepivacaine vs Bupivacaine Spinal Anesthesia for TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prisma Upstate
Record Dates: First submitted 2024-02-16; First posted 2024-03-04 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia, Spinal; Arthroplasty, Replacement, Knee
Keywords: knee arthroplasty; spinal anesthesia; same day discharge; mepivacaine; bupivacaine
MeSH Terms: interventions — Mepivacaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to one of two groups; one receiving Mepivacaine spinal anesthesia and the other receiving Bupivacaine spinal anesthesia for total knee arthroplasty (TKA).
Who Masked: Participant, Investigator
Masking Description: Investigators and participants will not know which anesthetic agent they receive. Anesthesia providers will be aware in order to provide correct randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepivacaine (Active Comparator): Standard dose of mepivacaine anesthesia (1.5% or 2%) for total knee arthroplasty procedure
  Interventions: Drug: Mepivacaine
- Bupivacaine (Active Comparator): Standard dose of hyperbaric bupivacaine anesthesia (0.75%) for total knee arthroplasty procedure
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Mepivacaine — Patients will be administered a standard dose of mepivacaine 1.5% (4.5ml, 67.5mg) for total knee arthroplasty prior to surgery
  Arms: Mepivacaine
Drug: Bupivacaine — Patients will be administered a standard dose of 0.75% hyperbaric bupivacaine (1.4ml, 10.5mg) for total knee arthroplasty prior to surgery
  Arms: Bupivacaine

SUMMARY:
This study is a prospective, double-blind prospective randomized controlled trial comparing mepivacaine and bupivacaine spinal anesthesia for same-day discharge readiness following a unilateral primary elective TKA procedure.

Study data will be collected during the patient's hospital stay for their TKA procedure, and the primary outcome of same-day discharge readiness will be assessed the day of surgery. Patients will also be contacted at Day 3 post-op to assess for any complications, current level of pain, and pain medication utilization.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the two different spinal anesthesia agents, mepivacaine and bupivacaine, and determine whether there are significant differences in their effects on readiness for same day discharge following a total knee arthroplasty.

This study is a prospective, double-blind prospective randomized controlled trial comparing mepivacaine and bupivacaine spinal anesthesia for same-day discharge readiness following a unilateral primary elective TKA procedure.

Study data will be collected during the patient's hospital stay for their TKA procedure, and the primary outcome of same-day discharge readiness will be assessed the day of surgery. Patients will also be contacted via telephone or RedCap at Day 3 post-op to assess for any complications, current level of pain, and pain medication utilization.

In this double-blind (patients and assessors) study, the patients will be randomly assigned 1:1 to receive one of the following: mepivacaine 1.5% (4.5ml, 67.5mg) or 2% (3.4ml, 67.5mg), (depending on availability from pharmacy) or hyperbaric bupivacaine 0.75% (1.4ml, 10.5mg) from the spinal kit. Randomization will be computer-generated in RedCap. These doses are the currently the standard doses used for our total knee arthroplasty patients. Patients with a height of 74 inches or greater or with body mass index of 35kg/m2 or greater will be given an extra 0.5ml of local anesthetic. The intraoperative anesthesia team will not be blinded to the group assignment, but patients, surgeons, and assessors are blinded. All patients will receive the standard preoperative multimodal analgesia, consisting of celecoxib 400mg po and acetaminophen 1gm po. Research staff will unblind the study investigators immediately if requested for any potential safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age who are scheduled for a primary elective TKA.
* Patient can ambulate at least 10 feet independently without human assistance.
* Patient must be a candidate for same day discharge as determined by American Society of Anesthesiologists (ASA) Physical Status Classification I and II

Exclusion Criteria:

* Patients scheduled for bilateral TKAs
* Contraindication to spinal anesthesia
* Revision TKAs
* Allergy or contraindication to NSAIDs (e.g. chronic anti-coagulant use)
* Workers' Compensation patient
* Type I Diabetes
* Type II Diabetes requiring insulin medication.
* Pre-operative narcotics use with the exception of tramadol.
* Renal insufficiency (GFR < 60) that may impact post-operative protocol
* Cognitive deficiencies that prevent the patient from providing their own informed consent
* Language barrier preventing completion of study forms in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Same day discharge rate | 24 hours
  Whether a patient is discharged the same day their surgery occurred, or if they were required to stay overnight following surgery.

SECONDARY OUTCOMES:
Post-operative pain score as assessed by numeric rating scale (NRS) | 3 days
  The NRS is a verbal pain scale that is evaluated on a scale of 0-10, with zero being no pain and 10 being 'the worst pain imaginable'. NRS pain scores will be collected while in the post-anesthesia care unit (PACU), at each physical therapy visit until discharge, and at 3 days post-operatively.
Urinary retention as assessed by time at which patient can voluntarily void bladder post-operatively | 24 hours
  Urinary retention will be evaluated based on whether patient is able to voluntarily void their bladder post-operatively. Time at which patient is able to voluntarily void their bladder will be recorded.
Return of sensory and motor function as assessed by ability of patient to plantar and dorsiflex lower extremity | 24 hours
  Time until return to sensory and motor function will be evaluated based on whether patient is able to plantar or dorsiflex lower extremity after surgery. Motor and sensory function will be considered 'intact' if patient is able perform these motions after surgery. Motor function will be evaluated in the post-anesthesia care unit (PACU) and during hospital stay over the course of 24 hours post-operatively.
Post-operative nausea and vomiting as assessed by clinical documentation of nausea and vomiting post-operatively | 24 hours
  Nausea and vomiting will be evaluated based on the presence of clinical documentation of episodes of nausea and vomiting during hospital admission over the course of 24 hours.
Pain Medications as evaluated by medical morphine equivalents | 24 hours
  Post-operative medications will be documented by medical morphine equivalents of medications administered during hospital stay. Total medical morphine equivalents over the course of 24 hours post-operatively will be used to capture pain medication usage during admission.
Patient satisfaction levels as assessed by a 5-item Likert response scale | 3 days
  Patient satisfaction levels will be captured using a 5-item Likert response scale with options of: 'very unsatisfied', 'unsatisfied', 'neutral', 'satisfied', and 'very satisfied' with respect to the type of anesthesia they received during their surgery. Satisfaction will be evaluated at Day 3 post-operative follow-up call.

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health Patewood Hospital, Greenville, South Carolina, United States